CLINICAL TRIAL: NCT01884623
Title: Multicentric Randomized Phase III Trial Comparing Methotrexate and Cetuximab in First-line Treatment of Recurrent and/or Metastatic Squamous Cell Head and Neck Cancer in Elderly Unfit Patients According to Geriatric Evaluation
Brief Title: Phase III Trial Comparing Methotrexate and Cetuximab in First-line Treatment of Recurrent and/or Metastatic Squamous Cell Head and Neck Cancer
Acronym: ELAN-UNFIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other); Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-004967-38; 2012/1937 (Other: CSET number)
Record Dates: First submitted 2013-06-18; First posted 2013-06-24 (Estimated); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Head Neck Cancer Squamous Cell Recurrent
MeSH Terms: interventions — Cetuximab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab (Experimental): Dosing schedule: 500 mg/m², every two weeks (q2w) Mode of administration: IV
  Interventions: Drug: Cetuximab
- Methotrexate (Active Comparator): Dosing schedule: 40mg/m2 weekly (q1w) Mode of administration: IV
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cetuximab
  Arms: Cetuximab
Drug: Methotrexate
  Arms: Methotrexate

SUMMARY:
To test whether cetuximab improves efficacy/tolerance as compared to methotrexate in first line treatment of unfit patients ³ 70 years old with recurrent and /or metastatic HNSCC. Efficacy assessed by failure free survival

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 70 or over
* Included in ELAN-ONCOVAL study and considered as "Unfit" by geriatric evaluation done in this study
* PS < 3
* Histologically confirmed diagnosis of squamous cell carcinoma of head and neck: oral cavity, oropharynx, hypopharynx, larynx.
* Recurrence and/or metastatic disease not suitable for local therapy.
* At least one measurable lesion (RECIST 1.1) by CT or MRI.
* No brain metastasis.
* Clearance of creatinine >= 50ml/mn (MDRD).
* Adequate haematological functions defined as follows: absolute neutrophil count > 1.5 x 109/l, platelet > 100 x 109/l, hemoglobin >= 9.5 g/dl
* Adequate hepatic functions with serum total bilirubin <1.25 Upper limit of normal range (ULN); SGOT/SGPT < 5 ULN; AP < 5 ULN
* Life expectancy > 12 weeks.
* Males of reproductive potential must agree to use an effective contraceptive method during the treatment and after the end of treatment during five months.
* Signed informed consent.
* Affiliated to Health Insurance regimen (according to Public Health Law of August 9, 2004).

Exclusion Criteria:

* Included in ELAN-ONCOVAL study and considered as "Fit" by geriatric evaluation
* Patients with nasopharyngeal cancer, paranasal sinus, or cervical lymph nodes metastasis of unknown origin.
* Prior systemic chemotherapy for the squamous cell carcinoma of head and neck, except if given as part of a multimodal treatment for locally advanced disease which was completed more than 6 months prior to study entry.
* Prior anti-EGFR therapy, except if given in association with radiotherapy for squamous cell carcinoma of head and neck which was completed more than 12 months prior to study entry.
* Surgery (excluding prior diagnostic biopsy) or irradiation within 4 weeks before study entry.
* Brain metastasis
* Active infection including tuberculosis and HIV infection.
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV), unstable angina pectoris, history of myocardial infarction within the last twelve months, significant arrhythmias
* Concomitant immunotherapy or antitumoral hormonotherapy.
* Requirement for treatment with any of the prohibited concomitant medications listed in SPC of Cetuximab and Methotrexate. In particular, acetylsalicylic acid used at analgesic, antipyretic or anti-inflammatory doses (see Section 6.3.2).
* Malignancies within 5 years prior to randomization, with the exception of adequately treated basal or squamous cell skin cancer and carcinoma in situ of the cervix
* Known allergic hypersensitivity to cetuximab or known positive results of tests for IgE antibodies against cetuximab (α-1-3-galactose) and/or methotrexate or any of their excipients.
* Other severe acute or chronic psychiatric or medical condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the patient's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Failure free survival (FFS) | From randomization to the first event among progression, treatment stop, whatever the cause, loss of 2 points or more in ADL scale and death assessed up to 16 months
  Composite criteria of efficacy and tolerance: Failure free survival (FFS) defined as time from randomization to the first event among progression (defined by RECIST criteria), treatment stop (whatever the cause), loss of 2 points or more in Activities in Daily Living (ADL) scale and death (whatever the cause). Patients who don't have any of these events are censored at the date of last follow-up.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause assessed up to 1 months
  Patients with disease progression will be treated off protocol but will be followed for overall survival evaluation.
Progression free survival (PFS) | From randomization to progression assessed up to 16 months
  minimum time from randomization to progression as defined by RECIST criteria or to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Joel GUIGAY, Pr, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Guigay J, Ortholan C, Vansteene D, Cupissol D, Even C, Kaminsky MC, Sire C, Blot E, Debourdeau P, Bozec L, Saada-Bouzid E, Fayette J, Dalloz P, Pointreau Y, Caer HL, Falandry C, Digue L, Braccini A, Lopez S, Guillet P, Michel C, Cheurfa N, Schwob D, Bourhis J, Mertens C, Auperin A; ELAN Group including Gustave Roussy, Unicancer GERICO and H&N groups and the GORTEC. Cetuximab versus methotrexate in first-line treatment of older, frail patients with inoperable recurrent or metastatic head and neck cancer (ELAN UNFIT): a randomised, open-label, phase 3 trial. Lancet Healthy Longev. 2024 Mar;5(3):e182-e193. doi: 10.1016/S2666-7568(23)00284-2. PMID 38432247